CLINICAL TRIAL: NCT04187937
Title: Feasibility of Ultrasound-based Navigation for Non-anatomical Liver Resections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruiting participants for the study due to the COVID-19 pandemic.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USGR
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Liver Neoplasm
Keywords: Image-Guidance; Liver Neoplasm
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-controlled, single-arm feasibility study of intraoperative ultrasound-based navigation for non-anatomical liver resections
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Stereotactic image-guided non-anatomical resection
  Interventions: Device: Stereotactic image-guided resection

INTERVENTIONS:
Device: Stereotactic image-guided resection — Stereotactic image-guided resection with an ultrasound-based image-guidance system.

SUMMARY:
In a non-anatomical resection of a liver tumor, only the part of the liver with the tumor and a safety margin of 5 - 10 mm are resected. This is done to ensure a negative resection margin, which means that no tumor cells are at the boundary of the resection. These non-anatomical resections can be performed repeatedly in case of recurrence. However, compared to anatomical resections, it is more challenging to keep a negative resection margin as anatomical landmarks cannot be used for intra-operative guidance.

In this study, the investigators aim to clinically evaluate a 3d navigation system, where navigated intra-operative ultrasound data is used to create a virtual model and a surgical plan.

DETAILED DESCRIPTION:
Surgical resection is the current gold standard for curative care of primary and metastatic hepatic tumors. This procedure involves the removal of the part of the liver where the tumor is located. This is typically achieved by removing the segments containing the tumor, so called anatomical resections. The downside of this technique is that it also removes a large part of healthy liver tissue. Recently, non-anatomical resections are becoming more popular, as they spare more healthy liver tissue than anatomical resections with similar oncological outcomes. In a non-anatomical resection, only the part of the liver with the tumor and a safety margin of 5 - 10 mm are resected. This is done to ensure a negative resection margin, which means that no tumor cells are at the boundary of the resection. These non-anatomical resections can be performed repeatedly in case of recurrence. However, compared to anatomical resections, it is more challenging to keep a negative resection margin as anatomical landmarks cannot be used for intra-operative guidance.

In the beginning of a non-anatomical resection, a resection line is drawn onto the liver surface to visualize where the resection shall be started. During the resection process, intra-operative ultrasound is used to confirm a safe distance to the tumor. Finally, once the depth is reached, the distance to the tumor is again confirmed on ultrasound and the tumor is removed. This is a challenging process which depends on the operator's ability and experience with mentally reconstructing the spatial relationships of the ultrasound image and the intra-operative scene. Additionally, the resection margin introduces artifacts and makes it harder to visualize the safety distance to the tumor on ultrasound.

To overcome these challenges, image-guidance systems have been introduced into the surgical workflow. These systems measure the pose of the surgical instruments and display their position on a virtual model of the anatomy. They mainly rely on a registration process to align a preoperative model with the patient's anatomy intraoperatively. This process is time-consuming, complex and error prone which is the main reason why such systems are rarely used.

In this study, the investigators aim to clinically evaluate a different approach, where navigated intra-operative ultrasound data is used to create a virtual model and a surgical plan on the spot. This does not require a separate registration process. With this approach a virtual draft of the surgical plan is created, which serves as a rough guidance map through the procedure. The investigators hypothesize that using such an intra-operative surgical draft allows the surgeon to acquire a negative resection margin.

ELIGIBILITY:
Inclusion Criteria:

* Patients which are regularly scheduled for an open surgical liver resection
* At least one tumor considered for non-anatomical resection
* Lesion is visible on ultrasound imaging
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age >= 18 years

Exclusion Criteria:

* Other clinically condition or disease that would (as deemed by the operating surgeon) significantly increase the risk of surgery
* Lesion is close to major vessel (< 10 mm)
* Lesion is too large to be visualized on ultrasound imaging
* Emergency
* Subjects not able to give informed consent (dementia)
* Women of childbearing potential (less than 1 year post-menopausal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 30 days
  Assessed by histopathological examination of the resected specimen. R0 is defined as a negative resection margin of >1 mm.

SECONDARY OUTCOMES:
Number of re-resections | intra-operative, expected to be up to 4 hours
Resection margin in mm | 30 days
Correlation with tumor size | pre-operative, expected to be up to 30 days
Correlation with tumor volume | pre-operative, expected to be up to 30 days
Correlation with tumor type | pre-operative, expected to be up to 30 days
Correlation with tumor location | pre-operative, expected to be up to 30 days
Time for planning of the resection | intra-operative, expected to be up to 4 hours
Time for resection | intra-operative, expected to be up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anja Lachenmayer, MD, Principal Investigator — Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Visceral Surgery and Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moris D, Tsilimigras DI, Kostakis ID, Ntanasis-Stathopoulos I, Shah KN, Felekouras E, Pawlik TM. Anatomic versus non-anatomic resection for hepatocellular carcinoma: A systematic review and meta-analysis. Eur J Surg Oncol. 2018 Jul;44(7):927-938. doi: 10.1016/j.ejso.2018.04.018. Epub 2018 Apr 30. PMID 29751946
- [Background] Banz VM, Muller PC, Tinguely P, Inderbitzin D, Ribes D, Peterhans M, Candinas D, Weber S. Intraoperative image-guided navigation system: development and applicability in 65 patients undergoing liver surgery. Langenbecks Arch Surg. 2016 Jun;401(4):495-502. doi: 10.1007/s00423-016-1417-0. Epub 2016 Apr 28. PMID 27122364
- [Background] Lango T, Vijayan S, Rethy A, Vapenstad C, Solberg OV, Marvik R, Johnsen G, Hernes TN. Navigated laparoscopic ultrasound in abdominal soft tissue surgery: technological overview and perspectives. Int J Comput Assist Radiol Surg. 2012 Jul;7(4):585-99. doi: 10.1007/s11548-011-0656-3. Epub 2011 Sep 3. PMID 21892604
- [Background] Kingham TP, Jayaraman S, Clements LW, Scherer MA, Stefansic JD, Jarnagin WR. Evolution of image-guided liver surgery: transition from open to laparoscopic procedures. J Gastrointest Surg. 2013 Jul;17(7):1274-82. doi: 10.1007/s11605-013-2214-5. Epub 2013 May 4. PMID 23645420